CLINICAL TRIAL: NCT05699239
Title: A Phase 2, Randomized, Placebo-controlled, Double-blind, Dose-finding Study of TS-172 in Hyperphosphatemia Patients on Hemodialysis
Brief Title: A Phase 2 Dose-finding Study of TS-172 in Hyperphosphatemia Patients on Hemodialysis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Taisho Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: TS172-02-01
Record Dates: First submitted 2023-01-12; First posted 2023-01-26 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2023-01

CONDITIONS: Hyperphosphatemia Patients on Hemodialysis
MeSH Terms: interventions — BID protein, human

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (5):
- 10 mg bid (Experimental): Patients receive TS-172 10 mg bid.
  Interventions: Drug: TS-172 10mg bid
- 30 mg bid (Experimental): Patients receive TS-172 30 mg bid.
  Interventions: Drug: TS-172 30mg bid
- 60 mg bid (Experimental): Patients receive TS-172 60 mg bid.
  Interventions: Drug: TS-172 60mg bid
- 20 mg tid (Experimental): Patients receive TS-172 20 mg tid.
  Interventions: Drug: TS-172 20mg tid
- Placebo (Placebo Comparator): Patients receive placebo.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: TS-172 10mg bid — oral administration of TS-172 10 mg bid
  Arms: 10 mg bid
Drug: TS-172 30mg bid — oral administration of TS-172 30 mg bid
  Arms: 30 mg bid
Drug: TS-172 60mg bid — oral administration of TS-172 60 mg bid
  Arms: 60 mg bid
Drug: TS-172 20mg tid — oral administration of TS-172 20 mg tid
  Arms: 20 mg tid
Drug: Placebo — oral administration of placebo
  Arms: Placebo

SUMMARY:
A phase 2, randomized, placebo-controlled, double-blind, dose-finding study of TS-172 in hyperphosphatemia patients on hemodialysis

ELIGIBILITY:
Inclusion Criteria:

1. Hyperphosphatemia patients (outpatients) with chronic kidney disease receiving hemodialysis (HD or HDF) 3 times a week for at least 12 weeks prior to Visit 1 (Week -4)
2. Patients aged ≥18 to <80 years at the time of obtaining informed consent
3. Patients with a serum phosphorus concentration of ≥ 3.5 mg/dL and ≤ 6.0 mg/dL at Visit 1 (Week -4)

Exclusion Criteria:

1. Patients with confirmed serum intact PTH concentration >500 pg/mL from Visit 1 (Week -4) to Visit 5 (Week 0)
2. Patients with serum phosphorus concentration ≥ 10.0 mg/dL from Visit 2 (Week -3) to Visit 5 (Week 0)
3. Patients who have undergone previous parathyroid intervention (PTx, PEIT, etc.)

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 326 (Actual)
Dates: Start 2023-02-08 (Actual); Primary Completion 2023-12-26 (Actual); Study Completion 2023-12-26 (Actual)

PRIMARY OUTCOMES:
Change from baseline in serum concentration of phosphorus | Week 4

SECONDARY OUTCOMES:
Achievement ratio of patients with the target serum concentration of phosphorus | Up to Week 4
Concentration of corrected serum calcium | Up to Week 4
Serum calcium times phosphorus product | Up to Week 4

CONTACTS AND LOCATIONS:
Overall Officials: Taisho Director, Study Director — Taisho Pharmaceutical Co., Ltd.
Locations (1):
- Taisho Pharmaceutical Co., Ltd selected site, Tokyo, Japan

IPD SHARING:
Plan to Share IPD: No